CLINICAL TRIAL: NCT03501381
Title: A Phase II Randomized, Open Label Study of High Dose Interleukin 2 vs High Dose Interleukin 2 Plus Entinostat in Advanced Renal Cell Carcinoma
Brief Title: High Dose IL 2 and Entinostat in RCC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roberto Pili (Other)
Collaborators: Indiana University Melvin and Bren Simon Cancer Center (Other); Syndax Pharmaceuticals (Industry); Clinigen, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Roberto Pili, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GU17-289
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — entinostat; Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- High Dose Interleukin 2 (Active Comparator): HD IL-2 600,000 IU/kg Every 8 hours on Days 1-5 and Days 15-19
  Interventions: Drug: Interleukin-2
- High Dose Interleukin 2 plus Entinostat (Experimental): HD IL-2 600,000 IU/kg Every 8 hours on Days 1-5 and Days 15-19 plus Entinostat 5 mg orally every 2 weeks starting Day -14
  Interventions: Drug: Entinostat; Drug: Interleukin-2

INTERVENTIONS:
Drug: Entinostat — Entinostat should be taken 1-2 hours prior to the HD IL-2 infusion. Dose reductions for entinostat should be followed. Entinostat will continue after high dose IL-2 every 2 weeks
  Arms: High Dose Interleukin 2 plus Entinostat
Drug: Interleukin-2 — In the event of clinical benefit after a course of HD IL-2 (stable disease or tumor shrinkage) patients will receive a second treatment course of HD IL-2 therapy. Patients with evidence of tumor shrinkage after the 2nd HD IL-2 treatment course may receive a 3rd treatment course of HD IL-2.
  Other Names: aldesleukin

SUMMARY:
This is a multicenter, randomized, open label study of high dose interleukin 2 vs high dose interleukin 2 plus entinostat in clear cell RCC patients who are candidate for high dose interleukin 2. Patients will be randomized to ARM 1 (high dose interleukin 2 plus entinostat) or ARM 2 (high dose interleukin 2). Subjects will receive up to 3 courses of high dose interleukin 600,000 units/kg administered IV every 8 hrs on Days 1-5 and Days 15-19 (maximum 28 doses) +/- entinostat 5 mg orally given every 2 weeks starting on Day-14, continuously. Tumor response assessment will be performed between HD IL-2 courses.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of 0 within 14 days prior to registration.
* Life expectancy of greater than 6 months.
* Patients must have pathological diagnosis of renal cell carcinoma that is metastatic or surgically unresectable. The histology must be clear cell carcinoma or predominant clear cell carcinoma.
* Patients must have measurable or evaluable disease by RECIST 1.1.
* Up to two prior therapies for RCC are allowed. One prior therapy must contain an immune checkpoint inhibitor.Prior palliative radiation to metastatic lesion(s) is permitted, provided there is at least one measurable and/or evaluable lesion(s) that has not been irradiated
* White blood cell (WBC) ≥ 3,000 K/mm3
* Absolute Neutrophil Count (ANC) ≥ 1,500/mm3
* Leukocytes ≥ 3,000/mm3
* Platelets ≥ 100,000/mm3
* Hemoglobin (Hgb) ≥ 12 g/dL
* Serum creatinine ≤ 1.5 x upper limit of normal (ULN)
* Calculated creatinine clearance ≥ 50 mL/min
* Corrected calcium ≤ 10 mg/dL
* Urine protein < 1 +; if ≥ 1+, a 24 hour urine protein should be obtained and be < 1,000 mg
* Total Bilirubin ≤ 1.5 × upper limit of normal (ULN)
* Aspartate aminotransferase (AST) ≤ 2.5 × ULN
* Alanine aminotransferase (ALT) ≤ 2.5 × ULN
* Lactate Dehydrogenase Within Normal Limits
* International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 × ULN
* Females of childbearing potential must have a negative serum pregnancy test during screening and within 3 days prior to receiving first dose of study medication. NOTE: Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.
* Females of childbearing potential and males must be willing to abstain from heterosexual activity or to use 2 forms of effective methods of contraception from the time of informed consent until 90days after treatment discontinuation. The two contraception methods can be comprised of two barrier methods, or a barrier method plus a hormonal method.
* Pulmonary: FEV1 > 2.0 liters or > 75% of predicted for height and age
* Cardiac: No evidence of congestive heart failure, symptoms of coronary artery disease, myocardial infarction less than 6 months prior to entry, serious cardiac arrhythmias, or unstable angina. NOTE: Patients who are over 40 or have had previous myocardial infarction greater than 6 months prior to entry will be required to have a negative or low probability cardiac stress test for cardiac ischemia.
* CNS: No history of cerebrovascular accident, transient ischemic attacks, central nervous system or brain metastases. NOTE: Patients with CNS metastases should have a head CT/MRI within 21 days prior to treatment initiation. Any imaging abnormality indicative of CNS metastases will exclude the patient from the study. Patients with previously excised/gamma knifed solitary or oligometastases and no evidence of recurrent disease for 6 months are eligible.

Exclusion Criteria:

* Prior treatment with HD IL-2
* Concurrent use of valproic acid use is not allowed.
* Receiving medications that can effect clotting ability: warfarin, aspirin (once-daily aspirin use- maximum dose 325 mg/day is permitted), nonsteroidal anti-inflammatory drugs (NSAIDs, including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents.
* Patients may not be receiving other investigational agents.
* Active infection requiring systemic therapy
* Pregnant or breastfeeding
* Any prior history of other cancer within the prior 5 years with the exception of adequately treated basal cell carcinoma, cervical intraepithelial neoplasia [CIN]/cervical carcinoma in situ, melanoma in situ or ductal carcinoma in situ [DCIS], localized Gleason 6 prostate cancer, papillary thyroid cancer or other non-melanoma skin cancers.
* Any medical condition that would preclude adequate evaluation of the safety and toxicity of the study combination.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure (New York Association Class II, III, or IV), angina pectoris requiring nitrate therapy, recent myocardial infarction (< the last 6 months), cardiac arrhythmia, history of CVA within 6 months, hypertension (defined as blood pressure of >160 mmHg systolic and/or >90 mmHg diastolic on medication), QTc interval > 470 msec, history of peripheral vascular disease, uncontrolled diabetes mellitus, or psychiatric illness/social situations that would limit compliance with study
* HIV-positive patients receiving combination antiretroviral therapy are are eligible if their HIV is well-controlled (undetectable VL and CD4 count >350) and they are on anti-retrovirals unlikely to interact with entinostat.
* Known active hepatitis B (e.g., hepatitis B surface antigen-reactive) or hepatitis C (e.g., hepatitis C virus ribonucleic acid [qualitative]). Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBc Ab] and absence of HBsAg) are eligible. NOTE: HBV DNA test must be performed prior to study treatment. Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Serious or non-healing wound, ulcer or bone fracture.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1 therapy.
* Anticipation of need for major surgical procedures during the course of the study.
* Left ventricular ejection function < 45%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2018-05-24 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 24 months
  Compare PFS between arms. PFS is defined as the time from date of randomization until the criteria for disease progression is met as defined by RECIST 1.1 or death as a result of any cause.

SECONDARY OUTCOMES:
Objective Response Rate | 24 months
  Estimate and compare the objective response rate in patients receiving high dose interleukin 2 or high dose interleukin 2 plus entinostat. ORR will include confirmed complete response (CR) + confirmed partial response (PR) and will be determined as per RECIST 1.1.
Assess Adverse Events | 24 months
  Assess the safety and tolerability of high dose interleukin 2 plus entinostat using CTCAE v4
Duration of response | 24 months
  Assess duration of response in patients receiving high dose interleukin 2 or high dose interleukin 2 plus entinostat. Duration of overall response-the period measured from the time that measurement criteria are met for complete or partial response (whichever status is recorded first) until the date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since treatment started).
Overall Survival | 24 Months
  Assess overall survival in patients receiving high dose interleukin 2 or high dose interleukin 2 plus entinostat. Overall survival is defined by the date of randomization to date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Pili, MD, Principal Investigator — Indiana University Melvin and Bren Simon Cancer Center
Locations (5):
- United States (5):
  - Univeristy of Southern California, Los Angeles, California
  - Rush University Medical Center, Chicago, Illinois
  - Indiana Univeristy Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Hematology Oncology Clinic, LLC, Baton Rouge, Louisiana
  - Nebraska Methodist Hospital, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: Undecided